CLINICAL TRIAL: NCT04118816
Title: Impact of Sleep-disordered Breathing on Autonomic Regulation in Patients With Prader-Willi Syndrome
Brief Title: Autonomic Regulation in Prader-Willi Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 08-XD-008
Record Dates: First submitted 2019-10-02; First posted 2019-10-08 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Autonomic Dysfunction
MeSH Terms: conditions — Primary Dysautonomias | interventions — Polysomnography; Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Healthy subjects, 7-75 y/o
  Interventions: Diagnostic Test: Polysomnography; Diagnostic Test: Multiple sleep latency test
- Study: 7-75 y/o, diagnosed with Prader-Willi syndrome.
  Interventions: Diagnostic Test: Polysomnography; Diagnostic Test: Multiple sleep latency test; Other: Continuous positive airway pressure

INTERVENTIONS:
Diagnostic Test: Polysomnography — overnight polysomnography recording at least six hours
  Other Names: PSG
Diagnostic Test: Multiple sleep latency test — daytime naps at least four to five naps to evaluate daytime sleepiness and narcolepsy
  Other Names: MSLT
Other: Continuous positive airway pressure — continuous positive airway pressure treatment for sleep-disordered breathing
  Other Names: CPAP
  Groups: Study

SUMMARY:
To evaluate autonomic regulation in patients with Prader-Willi syndrome with sleep-disordered breathing.

DETAILED DESCRIPTION:
To evaluate the relationship between narcolepsy and sleep-disordered breathing, the natural course of untreated or treated sleep-disordered breathing and its impacts on autonomic regulation in patients with Prader-Willi syndrome with sleep-disordered breathing.

ELIGIBILITY:
Inclusion Criteria:

* 7-75 y/o Prader-Willi syndrome patients or healthy subjects
* can perform polysomnography, multiple sleep latency test
* orthostatic methods for autonomic function test
* can perform pulmonary function test.

Exclusion Criteria:

* less than y/o, or larger then 75 y/o
* cannot perform polysomnography, multiple sleep latency test
* cannot orthostatic methods for autonomic function test
* cannot perform pulmonary function test
* use of sedatives or drugs affecting autonomic function

Ages: 7 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 7-75 y/o Prader-Willi syndrome patients or healthy subjects, can perform polysomnography, multiple sleep latency test, orthostatic methods for autonomic function test, can perform pulmonary function test.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-06-25 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Narcolepsy prevalence | 1day
  Compare the narcolepsy prevalence amount healthy and Prader-Willi syndrome with or without sleep-disordered breathing

SECONDARY OUTCOMES:
The natural course and its impact of untreated sleep-disordered breathing on autonomic regulation in patients with Prader-Willi syndrome. | 12 months
  Autonomic function measurements (low frequency power and high frequency power, presented as normalized units, and the overall autonomic regulation presented as Low frequency/high frequency ratio) using the EKG signal extracting from overnight polysomnography recording raw data among Prader-Willi patients with untreated sleep-disordered breathing at baseline and after a period of follow-up.

OTHER OUTCOMES:
The effect of continuous positive airway pressure on autonomic regulation in patients with Prader-Willi syndrome with sleep-disordered breathing. | 3 months
  1. Acute effect (one-night continuous positive airway pressure trial):
     Compared the autonomic function measurements between baseline polysomnography and one night continuous positive airway pressure treatment in patients with Prader-Willi Syndrome and sleep-disordered breathing.
  2. Chronic effect (at least 12 months treatment of continuous positive airway pressure) Compared the autonomic function measurements between baseline polysomnography and after at least 3 months continuous positive airway pressure treatment in patients with Prader-Willi Syndrome and sleep-disordered breathing.

CONTACTS AND LOCATIONS:
Overall Officials: 美貞 楊, MD, Principal Investigator — Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Locations (1):
- Taipei Tzu-Chi Hospital, Buddhist Tzu-Chi Medical Foundation, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghergan A, Coupaye M, Leu-Semenescu S, Attali V, Oppert JM, Arnulf I, Poitou C, Redolfi S. Prevalence and Phenotype of Sleep Disorders in 60 Adults With Prader-Willi Syndrome. Sleep. 2017 Dec 1;40(12). doi: 10.1093/sleep/zsx162. PMID 29294134
- [Background] Sedky K, Bennett DS, Pumariega A. Prader Willi syndrome and obstructive sleep apnea: co-occurrence in the pediatric population. J Clin Sleep Med. 2014 Apr 15;10(4):403-9. doi: 10.5664/jcsm.3616. PMID 24733986
- [Background] Miller J, Wagner M. Prader-Willi syndrome and sleep-disordered breathing. Pediatr Ann. 2013 Oct;42(10):200-4. doi: 10.3928/00904481-20130924-10. PMID 24126982
- [Background] Clift S, Dahlitz M, Parkes JD. Sleep apnoea in the Prader-Willi syndrome. J Sleep Res. 1994 Jun;3(2):121-126. doi: 10.1111/j.1365-2869.1994.tb00115.x. PMID 10607116
- [Background] Scammell TE. Narcolepsy. N Engl J Med. 2015 Dec 31;373(27):2654-62. doi: 10.1056/NEJMra1500587. No abstract available. PMID 26716917